CLINICAL TRIAL: NCT02613026
Title: Comparative Analysis of the Efficacies of AT and AC-T Regimens in Neoadjuvant Chemotherapy of Breast Cancer
Brief Title: Comparative Analysis of the Efficacies in Neoadjuvant Chemotherapy of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: 307 Hospital of PLA (Other)
Responsible Party: Principal Investigator, Shikai Wu, Chief Physician,Department of Radiotherapy, 307 Hospital of PLA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT2009
Record Dates: First submitted 2015-11-03; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Breast Neoplasms
Keywords: Breast tumor; Neoadjuvant chemotherapy; Pathological complete remission
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — pirarubicin; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined therapy group (Experimental): pirarubicin 50mg/m2, iv, d1; docetaxel 75mg/m2, div, d1. 21 days were a cycle of treatment, with a total of 4-8 cycles.
  Interventions: Drug: Pirarubicin; Drug: Docetaxel
- Sequential therapy group (Experimental): cyclophosphamide 600mg/m2, iv, d1; Pirarubicin 60mg/m2, iv, d1, 21 days were a cycle of treatment, with a total of 4 cycles. Then followed by Docetaxel 75- 100mg/m2, div, d1, 21 days were a cycle of treatment, with a total of 4 cycles.
  Interventions: Drug: Pirarubicin; Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pirarubicin
  Other Names: Tetrahydropyranyl Adriamycin
Drug: Docetaxel
  Other Names: Taxotere
Drug: Cyclophosphamide
  Arms: Sequential therapy group

SUMMARY:
The purpose of this study is to compare the short-term and long-term efficacies and the safeties of pirarubicin plus docetaxel(AT group) and pirarubicin plus cyclophosphamide followed by docetaxel(AC-T group) in neoadjuvant chemotherapy of breast cancer.

DETAILED DESCRIPTION:
Based on the results of NSABP(National Surgical Adjuvant Breast and Bowel Project) B27 trial, anthracyclines(A) and Taxanes(T) are most commonly recommended in neoadjuvant chemotherapy of breast cancer.

Pirarubicin is one of anthracyclines and by embedding the DNA double stranded, which inhibits DNA replication and RNA synthesis, thereby impedes the rapid growth of cancer cells.

Docetaxel in one of taxanes and by strengthening the tubulin polymerization, inhibiting of microtubule depolymerization and leading to the formation of stable non functional microtubule bundles, which destroys mitosis of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically diagnosed with stage I-III breast cancers;
* clearly confirmed ER, PR and HER2 statuses;
* the state of axillary lymph nodes was determined through the relevant examination steps (puncture or sentinel lymph node biopsy);
* the patients were not treated with neoadjuvant therapy and surgery.

Exclusion Criteria:

* the patients whose breasts or axillary lumps had received excision biopsy;
* the patients who had severely abnormal organ functions or who could not tolerate chemotherapy,
* the patients with severe concomitant diseases;
* the patients with heart disease or left ventricular ejection fraction (LVEF) <50%.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
pathological complete response rate | one year

SECONDARY OUTCOMES:
clinical response rate | one year
Percentage of changes in hormone receptors status after treatment | one year
Number of relative prognostic factors which influence pCR | three years

CONTACTS AND LOCATIONS:
Overall Officials: Shikai Wu, Principal Investigator — 307 Hospital of PLA
Locations (5):
- China (5):
  - The fourth hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

REFERENCES:
- [Background] Kaufmann M, Hortobagyi GN, Goldhirsch A, Scholl S, Makris A, Valagussa P, Blohmer JU, Eiermann W, Jackesz R, Jonat W, Lebeau A, Loibl S, Miller W, Seeber S, Semiglazov V, Smith R, Souchon R, Stearns V, Untch M, von Minckwitz G. Recommendations from an international expert panel on the use of neoadjuvant (primary) systemic treatment of operable breast cancer: an update. J Clin Oncol. 2006 Apr 20;24(12):1940-9. doi: 10.1200/JCO.2005.02.6187. PMID 16622270
- [Background] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Background] Mamounas EP, Brown A, Anderson S, Smith R, Julian T, Miller B, Bear HD, Caldwell CB, Walker AP, Mikkelson WM, Stauffer JS, Robidoux A, Theoret H, Soran A, Fisher B, Wickerham DL, Wolmark N. Sentinel node biopsy after neoadjuvant chemotherapy in breast cancer: results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2005 Apr 20;23(12):2694-702. doi: 10.1200/JCO.2005.05.188. PMID 15837984